CLINICAL TRIAL: NCT04091243
Title: Romosozumab Versus Denosumab for Osteoporosis in Long-term Glucocorticoid Users: an Open Randomized Controlled Trial
Brief Title: Romosozumab Versus Denosumab for Osteoporosis in Long-term Glucocorticoid Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTWC/REC/19074
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Glucocorticoid-induced Osteoporosis
Keywords: glucocorticoid; osteoporosis; rheumatic diseases
MeSH Terms: conditions — Osteoporosis; Rheumatic Diseases | interventions — romosozumab

STUDY DESIGN:
Intervention Model Description: An open randomized parallel group controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Romosozumab (Experimental): Romosozumab (210mg) subcutaneously every month for 12 doses
  Interventions: Drug: Romosozumab
- Denosumab (Active Comparator): Denosumab subcutaneously (60mg) every 6 months for 2 doses
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Experimental drug for the treatment of glucocorticoid induced osteoporosis

SUMMARY:
Glucocorticoid (GC) is the main stay of treatment of many rheumatic diseases but is also an important cause of secondary osteoporosis. The long-term use of GCs increases the risk of fragility fracture at a much higher bone mineral density (BMD) than postmenopausal osteoporosis, indicating an additional deleterious effect of GC on bone quality. An increased relative risk of vertebral and hip fractures is demonstrated in chronic GC users, with fracture risk proportional to the daily dose of GC. Other studies have also confirmed that intermittent use of high-dose GC and the cumulative GC dose was associated with an augmented risk of osteoporotic fracture.

Romosozumab (ROMO) is a humanized monoclonal antibody against sclerostin. The landmark RCT has demonstrated efficacy of ROMO (210mg subcutaneously monthly) over placebo in reducing vertebral fractures by 73% at 12 months in 7180 postmenopausal women with osteoporosis of the hip at entry. Another RCT has demonstrated efficacy of ROMO in reducing vertebral and hip fractures in 4093 post-menopausal women at month 24.

There are no data regarding the efficacy of ROMO in GC-induced osteoporosis. Comparative study on the efficacy of ROMO and denosumab in post-menopausal osteoporosis is also not yet available in the literature. This prompts the current pilot study to compare the efficacy of ROMO with denosumab in high-risk patients receiving long-term GCs.

DETAILED DESCRIPTION:
Glucocorticoid (GC) is the main stay of treatment of many rheumatic diseases but is also an important cause of secondary osteoporosis. The long-term use of GCs increases the risk of fragility fracture at a much higher bone mineral density (BMD) than postmenopausal osteoporosis, indicating an additional deleterious effect of GC on bone quality. More than one-third of postmenopausal women receiving GC therapy developed asymptomatic vertebral fractures. A study in general practice reported an increased relative risk of vertebral and hip fractures in chronic GC users, with fracture risk proportional to the daily dose of GC. Another study also confirmed that intermittent use of high-dose GC and the cumulative GC dose was associated with an augmented risk of osteoporotic fracture.

The glycoprotein sclerostin, secreted by the osteocytes under the influence of mechanical loading, inhibits activation of the canonical Wnt pathway involved in osteoblastogenesis and hence suppresses bone formation. Moreover, sclerostin enhances resorption of the bone by stimulating the production of (RANKL) by the osteocytes. Romosozumab (ROMO) is a humanized monoclonal antibody against sclerostin. The landmark RCT has demonstrated efficacy of ROMO (210mg subcutaneously monthly) over placebo in reducing vertebral fractures by 73% at 12 months in 7180 postmenopausal women with osteoporosis of the hip at entry. The suppression of markers of bone resorption and enhancement of markers of bone formation indicates that ROMO has a dual mode of action on the bones. The efficacy of ROMO has also been tested against oral bisphosphonates. A RCT was conducted in 4093 post-menopausal women who were assigned to receive either ROMO (201mg subcutaneously monthly) or oral alendronate (70mg weekly) for 12 months, followed by open-label alendronate for another 12 months. At month 24, a 48% lower risk of new vertebral fractures was observed in the ROMO (6.2%) than the alendronate group (11.9%; p<0.001). The risk of incident hip fractures was also significantly lower in the ROMO (2%) than alendronate treated patients (3.2%; p=0.02). The frequencies of adverse events and serious adverse events, however, were similar in the two treatment arms.

There are no data regarding the efficacy of ROMO in GC-induced osteoporosis. Comparative study on the efficacy of ROMO and denosumab in post-menopausal osteoporosis is also not yet available in the literature. This prompts the current pilot study to compare the efficacy of ROMO with denosumab in high-risk patients receiving long-term GCs.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (women or men) >18 years of age
2. Receiving long-term prednisolone treatment for various medical illnesses, defined as a daily prednisolone dose of ≥5mg/day for ≥12 months.
3. High risk of osteoporotic fracture (in subjects <40 years, personal history of fragility/vertebral fracture, bone mineral density [BMD] of the hip/spine Z score ≤ -3.0, loss of BMD >10% per year or new fracture; in subjects aged ≥40 years, personal history of fragility/vertebral fracture, BMD of the hip/spine T score ≤ -2.5, GC-adjusted 10-year major osteoporotic fracture risk ≥20% or hip fracture risk ≥3% by FRAX [ie. multiplying risk by 1.15 for the former and 1.20 for the latter when prednisolone ≥7.5mg/day], or new fracture development).

5. Informed consent from patients. 6. Willing to comply with all study procedures

Exclusion Criteria:

1. Patients with previous use of denosumab, teriparatide, intravenous bisphosphonates, strontium or other experimental anti-osteoporotic agents within 24 months of study entry.
2. Premenopausal women who plan for pregnancy within 24 months of study entry.
3. Patients with a known past history of atherosclerotic cardiovascular or cerebrovascular disease.
4. Patients with known bone disorders such as osteomalacia, renal osteodystrophy, and hyperparathyroidism.
5. Patients with unexplained hypocalcemia.
6. Patients with serum creatinine level of >=200umol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (BMD) | month 12
  Changes in BMD at lumbar spine from baseline

SECONDARY OUTCOMES:
Bone mineral density (BMD) | month 12
  Changes in BMD at the hip and femoral neck from baseline
bone turnover markers | months 6,12,18 and 24
  Changes in serum procollagen type 1 N-terminal propeptide (P1NP) and C-terminal telopeptide collagen degradation product of type 1 collagen (beta-CTX) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chi Chiu Mok, MD, FRCP, Principal Investigator — Tuen Mun Hospital
Locations (1):
- Tuen Mun Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No